CLINICAL TRIAL: NCT01086501
Title: Efficacy and Safety of an ER-formulation of Oxcarbazepine (Apydan Extent) in Epileptic Patients Under Consideration of Quality of Life Parameters
Brief Title: ESOXC-ER Efficacy and Safety of an Extended Release (ER) Formulation of Oxcarbazepine (Apydan Extent) in Epileptic Patients
Status: Completed | Type: Observational
Sponsor: Desitin Arzneimittel GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: OXC-044/K
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2010-03

CONDITIONS: Epilepsy
Keywords: open, non-interventional
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The aim of the observational study is to investigate the safety of oxcarbazepine extended release (ER) during long-term therapy in epileptic patients. In addition, quality of life parameters should be documented if assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients with focal epileptic seizures with or without secondary generalised tonic-clonic seizures
* mono- or combination therapy
* male and female from the age of 6

Exclusion Criteria:

* hypersensitivity to oxcarbazepine MR or one of its excipients

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: newly diagnosed epileptic patients or patients who will be switched from other antiepileptic drugs to oxcarbazepine ER
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2010-02; Primary Completion 2011-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
tolerability and safety | 12 months per patient

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Arnold, MD, Principal Investigator — Private Practice
Locations (1):
- Dr. Stephan Arnold, Munich, Bavaria, Germany

REFERENCES:
- [Background] Miller AD, Krauss GL, Hamzeh FM. Improved CNS tolerability following conversion from immediate- to extended-release carbamazepine. Acta Neurol Scand. 2004 Jun;109(6):374-7. doi: 10.1111/j.1600-0404.2004.00291.x. PMID 15147458